CLINICAL TRIAL: NCT02440126
Title: Longitudinal Meta-Analysis and Further Sample Collection To Evaluate Potential Host Markers for PML Risk
Brief Title: Longitudinal Analysis And Sample Collection To Evaluate PML Risk Host Markers for PML Risk Host Markers for PML Risk
Acronym: SRA-001
Status: Completed | Type: Observational
Sponsor: Rocky Mountain MS Research Group, LLC (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, John F. Foley, MD, President, Sponsor-Investigator, Rocky Mountain MS Research Group, LLC
Other Study IDs: SRA-001
Record Dates: First submitted 2014-10-16; First posted 2015-05-12 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; immunological; biomarkers; observational; Relapsing; Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group A: Natalizumab Naïve: This group will consist of up to 10 people who are naïve to natalizumab (haven't received the drug before) and are just beginning therapy. These participants will meet with the study staff at Week 0 (Baseline) prior to their natalizumab infusion. They will then have a follow up appointment every 3 months for the first 12 months of their natalizumab infusions, for a total of 5 visits. Natalizumab concentration and other biomarkers will be measured at each visit.
- Group B: Intracycle Regular Dosing: This group will consist of at least 50 people who are on a regular infusing cycle of 28-31 days. These participants will be consented at Week 0 (Baseline) and asked to come back each week during their regular cycle at Week 1, Week 2, and Week 3, for a total of 4 study visits. Natalizumab concentration and other biomarkers will be measured during their participation in the study.
- Group C: Intracycle Extended Dosing: This group will consist of up to 60 people who are on an extended infusing cycle of greater than 30 days. These participants will be consented at Week 0 (Baseline) and asked to come back each week for a blood draw to measure Natalizumab concentration and other biomarkers during their extended cycle at Week 2, and Week 4, for a total of 3 study visits.
- Group D: Transition Dosing: This group will consist of up to 10 people who are on a regular infusing cycle of 28-30 days who will be transitioning to an extended dosing cycle. The decision to transition will be made by their treating neurologist. These participants will be consented at Week 0 (Baseline) and will be followed for 8 cycles. Natalizumab concentration will be measured at each cycle. During certain cycles, other biomarkers will be measured.

SUMMARY:
The purpose of the study is to develop an improved understanding of the long term pharmacokinetics and pharmacodynamics of natalizumab with both standard dosing and extended dosing, and collect additional samples to explore cell-based biomarkers of natalizumab treatment and PML risk.

DETAILED DESCRIPTION:
The underlying etiology for the association of natalizumab therapy to an increase risk of progressive multifocal leukoencephalopathy (PML) remains unknown. It is possible that persistently high natalizumab levels lead to sustained immune-modulation or suppression resulting in an increased PML risk. Since 2010 we have conducted three investigator initiated trials (IITs) at our center to measure serum natalizumab concentration, lymphocyte alpha 4 integrin saturation, and other biomarkers to understand the association of these markers to PML risk. A number of the patients who participated in these clinical trials are still infusing. These studies have demonstrated that plasma natalizumab concentrations continue to rise over time with a plateau effect not yet clearly delineated. Improved drug clearance in patients with higher body weight is described in the prescribing information. We have accumulated preliminary data suggesting that patients with lower body weight may be at higher risk for PML and that this may relate to higher drug concentrations and saturations seen in this group. Dose extension may be a viable option to lower drug concentration (pharmacokinetic, PK) and saturation (pharmacodynamic, PD) in patients with lower body weight to potentially impact PML incidence. In addition to the PK/PD of natalizumab, host related biomarkers may allow for more specific PML risk stratification. Further validation of these biomarkers is critical for our understanding of their utility.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Must be enrolled in the TOUCH Prescribing Program for Tysabri® (natalizumab) prior to informed consent.
3. In the opinion of the Principal Investigator, must be able and willing to comply with all study directions
4. ≥ 18 years of age at the time of informed consent

Exclusion Criteria:

1. In the opinion of the Principal Investigator, subject is unwilling or unable to comply with study directions.
2. Subject who is pregnant, breastfeeding, or likely to becoming pregnant during the course of the study. Women of child-bearing potential must be practicing an acceptable form of birth control.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 patients with relapsing forms of multiple sclerosis. All subjects will receive open label natalizumab according to their prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Changes over Time | 12 month
  Changes in natalizumab concentration (ug/ml) will be collected and compared to similar infusion cycle lengths collected previously in investigator-initiated trials at this site.
Pharmacodynamic (PD) Changes over Time | 12 month
  Changes in natalizumab saturation (%) will be collected and compared to similar infusion cycle lengths collected previously in investigator-initiated trials at this site.

CONTACTS AND LOCATIONS:
Overall Officials: John F Foley, MD, Principal Investigator — Rocky Mountain MS Research Group, LLC
Locations (1):
- Rocky Mountain MS Research Group, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwab N, Schneider-Hohendorf T, Posevitz V, Breuer J, Gobel K, Windhagen S, Brochet B, Vermersch P, Lebrun-Frenay C, Posevitz-Fejfar A, Capra R, Imberti L, Straeten V, Haas J, Wildemann B, Havla J, Kumpfel T, Meinl I, Niessen K, Goelz S, Kleinschnitz C, Warnke C, Buck D, Gold R, Kieseier BC, Meuth SG, Foley J, Chan A, Brassat D, Wiendl H. L-selectin is a possible biomarker for individual PML risk in natalizumab-treated MS patients. Neurology. 2013 Sep 3;81(10):865-71. doi: 10.1212/WNL.0b013e3182a351fb. Epub 2013 Aug 7. PMID 23925765